CLINICAL TRIAL: NCT00005774
Title: Early Surfactant Followed by Nasal CPAP to Reduce the Use of Mechanical Ventilation Without Additional Morbidity in Infants 1250- 2000 Grams With RDS
Brief Title: Early Surfactant to Reduce Use of Mechanical Breathing in Low Birth Weight Infants
Acronym: Surfactant 2
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The trial was stopped after 7 months for lack of recruitment.
Sponsor: NICHD Neonatal Research Network (Network)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Responsible Party: Edward F. Donovan, Lead Principal Investigator, Cincinnati Children's Hospital Medical Center
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NICHD-NRN-0024; U10HD027856 (NIH); U10HD021364 (NIH); U10HD034216 (NIH); U10HD034167 (NIH); U10HD021397 (NIH); U10HD027853 (NIH); U10HD027871 (NIH); U10HD021415 (NIH); U10HD027904 (NIH); U10HD027881 (NIH); U10HD021385 (NIH); U10HD027851 (NIH); U10HD027880 (NIH); U01HD036790 (NIH); M01RR008084 (NIH); M01RR006022 (NIH); M01RR000750 (NIH); M01RR000997 (NIH); M01RR000070 (NIH); M01RR001032 (NIH)
Record Dates: First submitted 2000-06-01; First posted 2000-06-02 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Infant, Newborn; Respiratory Distress Syndrome; Respiratory Insufficiency
Keywords: NICHD Neonatal Research Network; Pulmonary ventilation; Respiratory distress syndrome; Respiratory insufficiency; Surfactant, pulmonary; Mechanical Ventilation; Survanta
MeSH Terms: conditions — Respiratory Distress Syndrome; Respiratory Insufficiency | interventions — beractant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early surfactant group (Experimental)
  Interventions: Drug: Early surfactant
- Standard Practice group (Active Comparator)
  Interventions: Drug: Standard practice

INTERVENTIONS:
Drug: Early surfactant — Early surfactant followed by extubation within 30 minutes and application of continuous positive airway pressure (CPAP)
  Other Names: Survanta
  Arms: Early surfactant group
Drug: Standard practice — Surfactant according to current center practice, only after initiation of mechanical ventilation.
  Arms: Standard Practice group

SUMMARY:
Mechanical ventilation (MV) of preterm infants with respiratory distress syndrome (RDS) is associated with lung injury and nosocomial infection. Moderately premature infants with mild respiratory distress do not routinely receive artificial surfactant early in their course of treatment. This multi-center, randomized trial tested whether early surfactant therapy and nasal continuous positive airway pressure (CPAP) in infants 1,250-2,000g with RDS reduced mechanical ventilation usage without added complications. Infants with mild to moderate respiratory distress syndrome were enrolled in the trial and given either early administration of surfactant followed by extubation within 30 minutes and the use of CPAP, or standard practice (surfactant according to current center practice, only after initiation of mechanical ventilation), to see whether the experimental method would reduce the need for subsequent mechanical ventilation.

DETAILED DESCRIPTION:
Mechanical ventilation (MV) of preterm infants with respiratory distress syndrome (RDS) is associated with lung injury and nosocomial infection. Moderately premature infants with mild respiratory distress do not routinely receive artificial surfactant early in their course of treatment. The role of surfactant therapy in the management of larger infants with respiratory distress syndrome (RDS) was unclear. In many neonatal intensive care units, these infants were routinely managed with continuous positive airway pressure (CPAP) alone.

This trial tested whether early use of surfactant combined with CPAP would ameliorate the course of RDS without an increased risk of death. Primary study outcomes were measures of use of mechanical ventilation, and thereby likely reduction in risk of ventilator-associated morbidity.

Eligible infants were randomized before the infant is 12 hours of age to receive either: early surfactant followed by extubation within 30 minutes and application of CPAP (intervention group); or surfactant according to current center practice, only after initiation of mechanical ventilation (control group).

The trial was stopped after 7 months for lack of recruitment.

ELIGIBILITY:
Inclusion Criteria:

* Infants born at 1,250-2g000 grams birth weight
* <12 hours of age
* Clinical and radiographic diagnosis of respiratory distress syndrome (RDS)
* Receiving supplemental oxygen with head-hood Fi02 of 0.35 to 0.50 or CPAP Fi02 of 0.25 to 0.50 to maintain oxygen saturation less than 90 percent and more than 96 percent

Exclusion Criteria:

* Receiving mechanical ventilation
* Air leak
* Pulmonary hemorrhage
* Major congenital anomaly
* Congenital non-bacterial infection
* Parental refusal of consent
* Refusal of attending neonatologist

Max Age: 12 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 61 (Actual)
Dates: Start 2000-05; Primary Completion 2002-07 (Actual); Study Completion 2002-07 (Actual)

PRIMARY OUTCOMES:
Need for mechanical ventilation following randomization | Until hospital discharge or 120 days of life

SECONDARY OUTCOMES:
Mean duration of mechanical ventilation | Until hospital discharge or 120 days of life
Risk morbidities associated with mechanical ventilation and/or early surfactant administration | Until hospital discharge or 120 days of life

CONTACTS AND LOCATIONS:
Overall Officials: Edward F. Donovan, MD, Study Director — Children's Hospital Medical Center, Cincinnati; David K. Stevenson, MD, Principal Investigator — Stanford University; Waldemar A. Carlo, MD, Principal Investigator — University of Alabama at Birmingham; Richard A. Ehrenkranz, MD, Principal Investigator — Yale University; Barbara J. Stoll, MD, Principal Investigator — Emory University; James A. Lemons, MD, Principal Investigator — Indiana University; Charles R. Bauer, MD, Principal Investigator — University of Miami; Lu-Ann Papile, MD, Principal Investigator — University of New Mexico; Seetha Shankaran, MD, Principal Investigator — Wayne State University; Avroy A. Fanaroff, MD, Principal Investigator — Case Western Reserve University, Rainbow Babies and Children's Hospital; William Oh, MD, Principal Investigator — Brown University, Women & Infants Hospital of Rhode Island; Sheldon B. Korones, MD, Principal Investigator — University of Tennessee; Jon E. Tyson, MD MPH, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (13):
- United States (13):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Stanford University, Palo Alto, California
  - Yale University, New Haven, Connecticut
  - University of Miami, Miami, Florida
  - Emory University, Atlanta, Georgia
  - Indiana University, Indianapolis, Indiana
  - Wayne State University, Detroit, Michigan
  - University of New Mexico, Albuquerque, New Mexico
  - Cincinnati Children's Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Brown University, Women & Infants Hospital of Rhode Island, Providence, Rhode Island
  - University of Tennessee, Memphis, Tennessee
  - University of Texas Health Science Center at Houston, Houston, Texas

REFERENCES:
- See also: NICHD Neonatal Research Network — http://neonatal.rti.org/